CLINICAL TRIAL: NCT03883412
Title: Effect of Exercise and/or Liraglutide on Vascular Dysfunction and Insulin Sensitivity in Type 2 Diabetes ( ZQL007)
Acronym: ZQL007
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: American Diabetes Association (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Zhenqi Liu, Professor and Chief, Division of Endocrinology and Metabolism, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20320
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Exercise; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Exercise Alone (Experimental): 16 weeks of treatment
  Interventions: Other: Exercise
- Liraglutide alone (Experimental): 16 weeks of treatment
  Interventions: Drug: Liraglutide
- Exercise + Liraglutide (Experimental): 16 weeks of treatment
  Interventions: Other: Exercise; Drug: Liraglutide

INTERVENTIONS:
Other: Exercise — 16 weeks of treatment
  Arms: Exercise + Liraglutide; Exercise Alone
Drug: Liraglutide — 16 weeks of Liraglutide
  Arms: Exercise + Liraglutide; Liraglutide alone

SUMMARY:
The primary objective of this study is to examine whether exercise training alone, liraglutide treatment alone or exercise training plus liraglutide treatment increases cardiac and muscle capillary blood volume, improves vascular function in the larger conduit vessels, and enhances insulin's metabolic action in humans with Type 2 diabetes. Subjects will be randomized to one of the three groups: exercise training, liraglutide treatment, and exercise + liraglutide. They will be studied at the baseline and then after 16 weeks of intervention.

DETAILED DESCRIPTION:
Our hypothesis is that sustained activation of the GLP-1 receptor with Liraglutide or exercise training will enhance microvascular perfusion, promote angiogenesis, and improve microvascular response to insulin in muscle, leading to increased muscle delivery of oxygen and nutrients and increased exercise tolerance in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60
* A1C ≤ 8.5%
* Never on GLP-1RA (eg: exenatide, liraglutide) or DPP4I ( eg: Sitaglipton)
* On stable dose of oral hypoglycemic agents >4 months
* On stable dose of other medications for >4 months

Exclusion Criteria:

* Taking Insulin
* Smoking presently or in the past 6 months
* BP >160/90
* BMI >35
* Family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome
* History of congestive heart failure, ischemic heart disease, severe pulmonary disease, liver or kidney disease.
* Any vascular disease such as myocardial infarction, stroke, peripheral vascular disease
* Presence of an intracardiac or intrapulmonary shunt (we will screen for this by auscultation during the physical exam by PI).
* Pregnant or breastfeeding.
* Known hypersensitivity to perflutren (contained in Definity)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Microvascular Blood Volume - change from baseline | 16 weeks
  measured at baseline and 16 weeks

SECONDARY OUTCOMES:
Augmentation Index - change from baseline | 16 weeks
  measured at baseline and 16 weeks
Flow Mediated Dilation - change from baseline | 16 weeks
  measured at baseline and 16 weeks
Pulse Wave Velocity - change from baseline | 16 weeks
  measured at baseline and 16 weeks
Post Ischemic Flow Velocity-Change from baseline | 16 weeks
  measured at baseline and 16 weeks
Insulin Sensitivity-Change from baseline | 16 weeks
  measured at baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhenqi Liu, MD, Principal Investigator — University of Virginia, Department of Endocrinoolgy
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamburg NM, Balady GJ. Exercise rehabilitation in peripheral artery disease: functional impact and mechanisms of benefits. Circulation. 2011 Jan 4;123(1):87-97. doi: 10.1161/CIRCULATIONAHA.109.881888. No abstract available. PMID 21200015
- [Background] Honig CR, Odoroff CL, Frierson JL. Active and passive capillary control in red muscle at rest and in exercise. Am J Physiol. 1982 Aug;243(2):H196-206. doi: 10.1152/ajpheart.1982.243.2.H196. PMID 7114231
- [Background] Barrett EJ, Eggleston EM, Inyard AC, Wang H, Li G, Chai W, Liu Z. The vascular actions of insulin control its delivery to muscle and regulate the rate-limiting step in skeletal muscle insulin action. Diabetologia. 2009 May;52(5):752-64. doi: 10.1007/s00125-009-1313-z. Epub 2009 Mar 13. PMID 19283361
- [Background] Vincent MA, Clerk LH, Lindner JR, Klibanov AL, Clark MG, Rattigan S, Barrett EJ. Microvascular recruitment is an early insulin effect that regulates skeletal muscle glucose uptake in vivo. Diabetes. 2004 Jun;53(6):1418-23. doi: 10.2337/diabetes.53.6.1418. PMID 15161743
- [Background] Eggleston EM, Jahn LA, Barrett EJ. Hyperinsulinemia rapidly increases human muscle microvascular perfusion but fails to increase muscle insulin clearance: evidence that a saturable process mediates muscle insulin uptake. Diabetes. 2007 Dec;56(12):2958-63. doi: 10.2337/db07-0670. Epub 2007 Aug 24. PMID 17720897
- [Background] Chai W, Wang W, Liu J, Barrett EJ, Carey RM, Cao W, Liu Z. Angiotensin II type 1 and type 2 receptors regulate basal skeletal muscle microvascular volume and glucose use. Hypertension. 2010 Feb;55(2):523-30. doi: 10.1161/HYPERTENSIONAHA.109.145409. Epub 2009 Dec 7. PMID 19996061
- [Background] Liu Z, Liu J, Jahn LA, Fowler DE, Barrett EJ. Infusing lipid raises plasma free fatty acids and induces insulin resistance in muscle microvasculature. J Clin Endocrinol Metab. 2009 Sep;94(9):3543-9. doi: 10.1210/jc.2009-0027. Epub 2009 Jun 30. PMID 19567533
- [Background] Liu J, Jahn LA, Fowler DE, Barrett EJ, Cao W, Liu Z. Free fatty acids induce insulin resistance in both cardiac and skeletal muscle microvasculature in humans. J Clin Endocrinol Metab. 2011 Feb;96(2):438-46. doi: 10.1210/jc.2010-1174. Epub 2010 Nov 3. PMID 21047922
- [Background] Vincent MA, Barrett EJ, Lindner JR, Clark MG, Rattigan S. Inhibiting NOS blocks microvascular recruitment and blunts muscle glucose uptake in response to insulin. Am J Physiol Endocrinol Metab. 2003 Jul;285(1):E123-9. doi: 10.1152/ajpendo.00021.2003. PMID 12791603
- [Background] Jiang ZY, Lin YW, Clemont A, Feener EP, Hein KD, Igarashi M, Yamauchi T, White MF, King GL. Characterization of selective resistance to insulin signaling in the vasculature of obese Zucker (fa/fa) rats. J Clin Invest. 1999 Aug;104(4):447-57. doi: 10.1172/JCI5971. PMID 10449437
- [Background] Kim JA, Koh KK, Quon MJ. The union of vascular and metabolic actions of insulin in sickness and in health. Arterioscler Thromb Vasc Biol. 2005 May;25(5):889-91. doi: 10.1161/01.ATV.0000164044.42910.6b. No abstract available. PMID 15863720
- [Background] Kim JA, Montagnani M, Koh KK, Quon MJ. Reciprocal relationships between insulin resistance and endothelial dysfunction: molecular and pathophysiological mechanisms. Circulation. 2006 Apr 18;113(15):1888-904. doi: 10.1161/CIRCULATIONAHA.105.563213. PMID 16618833
- [Background] Rattigan S, Clark MG, Barrett EJ. Acute vasoconstriction-induced insulin resistance in rat muscle in vivo. Diabetes. 1999 Mar;48(3):564-9. doi: 10.2337/diabetes.48.3.564. PMID 10078557
- [Background] Youd JM, Rattigan S, Clark MG. Acute impairment of insulin-mediated capillary recruitment and glucose uptake in rat skeletal muscle in vivo by TNF-alpha. Diabetes. 2000 Nov;49(11):1904-9. doi: 10.2337/diabetes.49.11.1904. PMID 11078458
- [Background] Clerk LH, Rattigan S, Clark MG. Lipid infusion impairs physiologic insulin-mediated capillary recruitment and muscle glucose uptake in vivo. Diabetes. 2002 Apr;51(4):1138-45. doi: 10.2337/diabetes.51.4.1138. PMID 11916937
- [Background] Wallis MG, Wheatley CM, Rattigan S, Barrett EJ, Clark AD, Clark MG. Insulin-mediated hemodynamic changes are impaired in muscle of Zucker obese rats. Diabetes. 2002 Dec;51(12):3492-8. doi: 10.2337/diabetes.51.12.3492. PMID 12453905
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Chai W, Liu J, Jahn LA, Fowler DE, Barrett EJ, Liu Z. Salsalate attenuates free fatty acid-induced microvascular and metabolic insulin resistance in humans. Diabetes Care. 2011 Jul;34(7):1634-8. doi: 10.2337/dc10-2345. Epub 2011 May 26. PMID 21617098
- [Background] Potenza MA, Marasciulo FL, Chieppa DM, Brigiani GS, Formoso G, Quon MJ, Montagnani M. Insulin resistance in spontaneously hypertensive rats is associated with endothelial dysfunction characterized by imbalance between NO and ET-1 production. Am J Physiol Heart Circ Physiol. 2005 Aug;289(2):H813-22. doi: 10.1152/ajpheart.00092.2005. Epub 2005 Mar 25. PMID 15792994
- [Background] Eringa EC, Stehouwer CD, Merlijn T, Westerhof N, Sipkema P. Physiological concentrations of insulin induce endothelin-mediated vasoconstriction during inhibition of NOS or PI3-kinase in skeletal muscle arterioles. Cardiovasc Res. 2002 Dec;56(3):464-71. doi: 10.1016/s0008-6363(02)00593-x. PMID 12445887
- [Background] Eringa EC, Stehouwer CD, van Nieuw Amerongen GP, Ouwehand L, Westerhof N, Sipkema P. Vasoconstrictor effects of insulin in skeletal muscle arterioles are mediated by ERK1/2 activation in endothelium. Am J Physiol Heart Circ Physiol. 2004 Nov;287(5):H2043-8. doi: 10.1152/ajpheart.00067.2004. Epub 2004 Apr 1. PMID 15059773
- [Background] Lillioja S, Young AA, Culter CL, Ivy JL, Abbott WG, Zawadzki JK, Yki-Jarvinen H, Christin L, Secomb TW, Bogardus C. Skeletal muscle capillary density and fiber type are possible determinants of in vivo insulin resistance in man. J Clin Invest. 1987 Aug;80(2):415-24. doi: 10.1172/JCI113088. PMID 3301899
- [Background] Gavin TP, Stallings HW 3rd, Zwetsloot KA, Westerkamp LM, Ryan NA, Moore RA, Pofahl WE, Hickner RC. Lower capillary density but no difference in VEGF expression in obese vs. lean young skeletal muscle in humans. J Appl Physiol (1985). 2005 Jan;98(1):315-21. doi: 10.1152/japplphysiol.00353.2004. Epub 2004 Aug 6. PMID 15298982
- [Background] Akerstrom T, Laub L, Vedel K, Brand CL, Pedersen BK, Lindqvist AK, Wojtaszewski JF, Hellsten Y. Increased skeletal muscle capillarization enhances insulin sensitivity. Am J Physiol Endocrinol Metab. 2014 Dec 15;307(12):E1105-16. doi: 10.1152/ajpendo.00020.2014. Epub 2014 Oct 28. PMID 25352432
- [Background] Olsson AK, Dimberg A, Kreuger J, Claesson-Welsh L. VEGF receptor signalling - in control of vascular function. Nat Rev Mol Cell Biol. 2006 May;7(5):359-71. doi: 10.1038/nrm1911. PMID 16633338
- [Background] Hazarika S, Dokun AO, Li Y, Popel AS, Kontos CD, Annex BH. Impaired angiogenesis after hindlimb ischemia in type 2 diabetes mellitus: differential regulation of vascular endothelial growth factor receptor 1 and soluble vascular endothelial growth factor receptor 1. Circ Res. 2007 Oct 26;101(9):948-56. doi: 10.1161/CIRCRESAHA.107.160630. Epub 2007 Sep 6. PMID 17823371
- [Background] Tang K, Breen EC, Gerber HP, Ferrara NM, Wagner PD. Capillary regression in vascular endothelial growth factor-deficient skeletal muscle. Physiol Genomics. 2004 Jun 17;18(1):63-9. doi: 10.1152/physiolgenomics.00023.2004. Epub 2004 Jun 17. PMID 15084712
- [Background] Bonner JS, Lantier L, Hasenour CM, James FD, Bracy DP, Wasserman DH. Muscle-specific vascular endothelial growth factor deletion induces muscle capillary rarefaction creating muscle insulin resistance. Diabetes. 2013 Feb;62(2):572-80. doi: 10.2337/db12-0354. Epub 2012 Sep 21. PMID 23002035
- [Background] Robbins JL, Jones WS, Duscha BD, Allen JD, Kraus WE, Regensteiner JG, Hiatt WR, Annex BH. Relationship between leg muscle capillary density and peak hyperemic blood flow with endurance capacity in peripheral artery disease. J Appl Physiol (1985). 2011 Jul;111(1):81-6. doi: 10.1152/japplphysiol.00141.2011. Epub 2011 Apr 21. PMID 21512146
- [Background] Lindner JR, Womack L, Barrett EJ, Weltman J, Price W, Harthun NL, Kaul S, Patrie JT. Limb stress-rest perfusion imaging with contrast ultrasound for the assessment of peripheral arterial disease severity. JACC Cardiovasc Imaging. 2008 May;1(3):343-50. doi: 10.1016/j.jcmg.2008.04.001. PMID 19356447
- [Background] Hiatt WR, Wolfel EE, Meier RH, Regensteiner JG. Superiority of treadmill walking exercise versus strength training for patients with peripheral arterial disease. Implications for the mechanism of the training response. Circulation. 1994 Oct;90(4):1866-74. doi: 10.1161/01.cir.90.4.1866. PMID 7923674
- [Background] Brendle DC, Joseph LJ, Corretti MC, Gardner AW, Katzel LI. Effects of exercise rehabilitation on endothelial reactivity in older patients with peripheral arterial disease. Am J Cardiol. 2001 Feb 1;87(3):324-9. doi: 10.1016/s0002-9149(00)01367-9. PMID 11165969
- [Background] Schlager O, Giurgea A, Schuhfried O, Seidinger D, Hammer A, Groger M, Fialka-Moser V, Gschwandtner M, Koppensteiner R, Steiner S. Exercise training increases endothelial progenitor cells and decreases asymmetric dimethylarginine in peripheral arterial disease: a randomized controlled trial. Atherosclerosis. 2011 Jul;217(1):240-8. doi: 10.1016/j.atherosclerosis.2011.03.018. Epub 2011 Apr 8. PMID 21481871
- [Background] Januszek R, Mika P, Konik A, Petriczek T, Nowobilski R, Nizankowski R. Effect of treadmill training on endothelial function and walking abilities in patients with peripheral arterial disease. J Cardiol. 2014 Aug;64(2):145-51. doi: 10.1016/j.jjcc.2013.12.002. Epub 2014 Jan 14. PMID 24438856
- [Background] Ernst EE, Matrai A. Intermittent claudication, exercise, and blood rheology. Circulation. 1987 Nov;76(5):1110-4. doi: 10.1161/01.cir.76.5.1110. PMID 3499255
- [Background] Vincent MA, Clerk LH, Lindner JR, Price WJ, Jahn LA, Leong-Poi H, Barrett EJ. Mixed meal and light exercise each recruit muscle capillaries in healthy humans. Am J Physiol Endocrinol Metab. 2006 Jun;290(6):E1191-7. doi: 10.1152/ajpendo.00497.2005. PMID 16682488
- [Background] Hoier B, Hellsten Y. Exercise-induced capillary growth in human skeletal muscle and the dynamics of VEGF. Microcirculation. 2014 May;21(4):301-14. doi: 10.1111/micc.12117. PMID 24450403
- [Background] Inyard AC, Clerk LH, Vincent MA, Barrett EJ. Contraction stimulates nitric oxide independent microvascular recruitment and increases muscle insulin uptake. Diabetes. 2007 Sep;56(9):2194-200. doi: 10.2337/db07-0020. Epub 2007 Jun 11. PMID 17563063
- [Background] Wheatley CM, Rattigan S, Richards SM, Barrett EJ, Clark MG. Skeletal muscle contraction stimulates capillary recruitment and glucose uptake in insulin-resistant obese Zucker rats. Am J Physiol Endocrinol Metab. 2004 Oct;287(4):E804-9. doi: 10.1152/ajpendo.00077.2004. Epub 2004 Jun 22. PMID 15213062
- [Background] St-Pierre P, Keith LJ, Richards SM, Rattigan S, Keske MA. Microvascular blood flow responses to muscle contraction are not altered by high-fat feeding in rats. Diabetes Obes Metab. 2012 Aug;14(8):753-61. doi: 10.1111/j.1463-1326.2012.01598.x. Epub 2012 Apr 18. PMID 22429614
- [Background] Olfert IM, Howlett RA, Tang K, Dalton ND, Gu Y, Peterson KL, Wagner PD, Breen EC. Muscle-specific VEGF deficiency greatly reduces exercise endurance in mice. J Physiol. 2009 Apr 15;587(Pt 8):1755-67. doi: 10.1113/jphysiol.2008.164384. Epub 2009 Feb 23. PMID 19237429
- [Background] Stevens JW, Simpson E, Harnan S, Squires H, Meng Y, Thomas S, Michaels J, Stansby G. Systematic review of the efficacy of cilostazol, naftidrofuryl oxalate and pentoxifylline for the treatment of intermittent claudication. Br J Surg. 2012 Dec;99(12):1630-8. doi: 10.1002/bjs.8895. Epub 2012 Oct 3. PMID 23034699
- [Background] Fakhry F, van de Luijtgaarden KM, Bax L, den Hoed PT, Hunink MG, Rouwet EV, Spronk S. Supervised walking therapy in patients with intermittent claudication. J Vasc Surg. 2012 Oct;56(4):1132-42. doi: 10.1016/j.jvs.2012.04.046. PMID 23026425
- [Background] Zhao T, Parikh P, Bhashyam S, Bolukoglu H, Poornima I, Shen YT, Shannon RP. Direct effects of glucagon-like peptide-1 on myocardial contractility and glucose uptake in normal and postischemic isolated rat hearts. J Pharmacol Exp Ther. 2006 Jun;317(3):1106-13. doi: 10.1124/jpet.106.100982. Epub 2006 Feb 17. PMID 16489128